CLINICAL TRIAL: NCT05032742
Title: Reducing Parenting Stress to Facilitate Justice-Involved Youth's Treatment
Brief Title: Parenting Stress mHealth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: K23DA050798 (NIH); K23DA050798 (NIH)
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Stress
Keywords: parenting stress; juvenile justice; digital health

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth parenting stress app (Experimental): mHealth parenting stress app intervention to reduce parenting stress and improving youth community-based treatment engagement.
  Interventions: Behavioral: mHealth parenting stress app
- Standard of care (No Intervention): Caregiver participants will receive an informational brochure describing ways to support one's adolescent during detention and community reentry and any other usual care.

INTERVENTIONS:
Behavioral: mHealth parenting stress app — mHealth parenting stress app intervention to reduce parenting stress and improving youth community-based treatment engagement.
  Arms: mHealth parenting stress app

SUMMARY:
Parenting stress is a well-documented barrier to youth engagement in community-based substance use treatment. The current project aims to develop and evaluate a mobile health parenting stress intervention for caregivers of justice-involved youth, a population with high rates of substance use and low rates of treatment engagement.

DETAILED DESCRIPTION:
Justice-involved youth exhibit high rates of substance use and mental health symptoms, yet few receive treatment during detention or community re-entry. Once released into the community, caregivers must facilitate youth's treatment engagement, mobilizing significant resources and facing many barriers (e.g., transportation, mistrust) to do so. Parenting stress, which is heightened during youth detention and community reentry, is associated with greater perceived barriers to treatment, less youth therapeutic change throughout treatment, and premature treatment dropout. Addressing parenting stress improves youth treatment engagement and outcomes among youth exhibiting antisocial behavior, yet given the many barriers to treatment, novel approaches to intervention are needed; mobile health (mHealth) technology is one promising approach. Caregivers of justice-involved youth and system stakeholders are interested in mHealth treatment and mHealth addresses instrumental barriers (e.g., transportation) to treatment. Advances in technology and community engaged research allow for active stakeholder collaboration in mHealth application development, with no technological expertise required, through participatory informatics; caregiver involvement increases the likelihood the intervention will be relevant and efficacious. The purpose of this mixed-methods K23 study is to 1) develop a mHealth parenting stress intervention using participatory informatics; 2) assess the feasibility and acceptability of the participatory informatics approach and the intervention; 3) evaluate the intervention's preliminary efficacy in reducing parenting stress and increasing youth engagement in substance use or dual diagnosis treatment post-detention through a pilot randomized controlled trial; and 4) understand systems-level factors that could influence eventual system adoption and sustainability.

ELIGIBILITY:
Inclusion Criteria:

The following is a description for the inclusion criteria for aims 1 and 2 for caregivers participating in this research study.

Eligible caregivers must be the parent or legal guardian of a youth who is:

* currently detained in a juvenile detention center or correctional facility, mandated by the juvenile justice system to a congregate out-of-home placement (e.g., group home);
* 12-17 years old;
* has an identified substance use or substance use and co-occurring mental health need;
* and is scheduled to be released into the community to the care of the enrolled caregiver.

The following is a description for the inclusion criteria for aim 3 for system stakeholders participating in this research study.

Eligible behavioral health providers (e.g., substance use counselor) must:

* Provide substance use or dual diagnosis treatment justice-involved youth and their caregivers,
* be over 18 years old,
* and speak English fluently.

Eligible juvenile probation officers must be:

* 18 years or older
* and speak fluent English.

Exclusion Criteria:

Exclusion criteria for all participants includes:

* lack of proficiency in English
* and cognitive impairment or active psychosis which precludes provision of informed consent.

Caregivers who do not have access to a device with internet access will also not be eligible as this would preclude them from being able to participate in the mHealth intervention.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Interpersonal Mindfulness in Parenting Scale (Mindful Parenting) | 3 months post baseline
  The Interpersonal Mindfulness in Parenting Scale is an 8-item self-report of mindful parenting, including four sub-scales reflecting present-centered emotional awareness in parenting, present-centered attention in parenting, non-reactivity/low reactivity in parenting, and non-judgmental acceptance in parenting that will be used to measure mindful parenting as a construct. Each item is rated on a 1 to 5 scale and items are summed to create sub-scale scores (possible range=8 to 40); higher scores indicate greater mindful parenting.
Interpersonal Mindfulness in Parenting Scale (Mindful Parenting) | 6 months post baseline
  The Interpersonal Mindfulness in Parenting Scale is an 8-item self-report of mindful parenting, including four sub-scales reflecting present-centered emotional awareness in parenting, present-centered attention in parenting, non-reactivity/low reactivity in parenting, and non-judgmental acceptance in parenting that will be used to measure mindful parenting as a construct. Each item is rated on a 1 to 5 scale and items are summed to create sub-scale scores (possible range=8 to 40); higher scores indicate greater mindful parenting.
Stress Index for Parents of Adolescents (Parenting Stress) | 3 months post baseline
  The Stress Index for Parents of Adolescents (SIPA) is a 90-item self-report measure of parenting stress. Items are rated on a 1 to 5 scale and summed to create sub-scale scores; higher scores reflect greater parenting stress.
Stress Index for Parents of Adolescents (Parenting Stress) | 6 months post baseline
  The Stress Index for Parents of Adolescents (SIPA) is a 90-item self-report measure of parenting stress. Items are rated on a 1 to 5 scale and summed to create sub-scale scores (possible range=90 to 450); higher scores reflect greater parenting stress.
Parenting Self-Efficacy | 3 months post baseline
  Parenting Self-Efficacy Scale (PSES) is a 20-item assessment of caregivers' perceived parenting ability across 3 dimensions: parental connection, behavioral influence, and psychological autonomy and used to measure parenting self-efficacy. Items are rated on a scale from 0 to 10 (possible range=0 to 200) with higher scores reflecting greater parenting self-efficacy.
Parenting Self-Efficacy | 6 months post baseline
  Parenting Self-Efficacy Scale (PSES) is a 20-item assessment of caregivers' perceived parenting ability across 3 dimensions: parental connection, behavioral influence, and psychological autonomy and used to measure parenting self-efficacy. Items are rated on a scale from 0 to 10 (possible range=0 to 200) with higher scores reflecting greater parenting self-efficacy.
Child and Adolescent Services Assessment (Barriers to Youth Treatment) | 3 months post baseline
  The Child and Adolescent Services Assessment (CASA) is a parent-report instrument designed to assess the use of behavioral health services by children ages 8 years to 17 years. The CASA includes 31 settings covering inpatient, outpatient, and informal services provided by a variety of child-serving providers and sectors. This instrument collects information on whether a service was ever used, as well as more detailed information (length of stay/number of visits, focus of treatment) on services used in the recent past. Select items from the CASA will assess 16 barriers to youths' services use (e.g., language, transportation, cost, stigma). Caregivers will report whether each barrier was a concern during the 3 months prior to the youths' detention or for follow-ups, in the 3 months since the last assessment (6 months post baseline).
Child and Adolescent Services Assessment (Barriers to Youth Treatment) | 6 months post baseline
  The Child and Adolescent Services Assessment (CASA) is a parent-report instrument designed to assess the use of behavioral health services by children ages 8 years to 17 years. The CASA includes 31 settings covering inpatient, outpatient, and informal services provided by a variety of child-serving providers and sectors. This instrument collects information on whether a service was ever used, as well as more detailed information (length of stay/number of visits, focus of treatment) on services used in the recent past. Select items from the CASA will assess 16 barriers to youths' services use (e.g., language, transportation, cost, stigma). Caregivers will report whether each barrier was a concern during the 3 months prior to the youths' detention or for follow-ups, in the 3 months since the last assessment (6 months post baseline).
Motivation for Youth Treatment | 3 months post baseline
  Motivation for Youth's Treatment Scale (MYTS) is an 8-item measure of intrinsic motivation for youth treatment and assesses a youth and caregiver's problem recognition and treatment readiness. Responses are rated on a 1 to 5 scale and are summed to yield two sub-scale scores (problem recognition: possible range=3 to 15; treatment readiness: possible range=5 to 25). Higher scores reflect higher motivation.
Motivation for Youth Treatment | 6 months post baseline
  Motivation for Youth's Treatment Scale (MYTS) is an 8-item measure of intrinsic motivation for youth treatment and assesses a youth and caregiver's problem recognition and treatment readiness. Responses are rated on a 1 to 5 scale and are summed to yield two sub-scale scores (problem recognition: possible range=3 to 15; treatment readiness: possible range=5 to 25). Higher scores reflect higher motivation.

SECONDARY OUTCOMES:
Youth Treatment Engagement | 3 months post baseline
  Caregiver report on whether youth initiated substance use, mental health, dual diagnosis, or family based treatment in the community (i.e., scheduled appointment, attended first appointment), treatment retention (i.e., number of sessions attended) is collected to measure youth treatment engagement. Caregiver report will also provide information on whether the youth complied with treatment mandated by the juvenile court (e.g., probation requirement).
Youth Treatment Engagement | 6 months post baseline
  Caregiver report on whether youth initiated substance use, mental health, dual diagnosis, or family based treatment in the community (i.e., scheduled appointment, attended first appointment), treatment retention (i.e., number of sessions attended) is collected to measure youth treatment engagement. Caregiver report will also provide information on whether the youth complied with treatment mandated by the juvenile court (e.g., probation requirement).

OTHER OUTCOMES:
Caregiver Mental Health & Substance Use | 3 months post baseline
  Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) Cross Cutting Symptom Inventory is a 23-item self-report assessment of psychiatric symptoms (e.g., depression, anxiety, mania, psychosis) and substance use during the past 2 weeks; 1 item regarding suicidal ideation was removed. Items are rated on a scale from 0 to 4 (possible range=0 to 88). Higher scores reflect greater symptom severity.
Caregiver Mental Health & Substance Use | 6 months post baseline
  DSM-5 Cross Cutting Symptom Inventory is a 23-item self-report assessment of psychiatric symptoms (e.g., depression, anxiety, mania, psychosis) and substance use during the past 2 weeks; 1 item regarding suicidal ideation was removed. Items are rated on a scale from 0 to 4 (possible range=0 to 88). Higher scores reflect greater symptom severity.
mHealth Application Acceptability | 3 months post baseline
  Completed by the intervention condition only, the mHealth App Usability Questionnaire for Standalone mHealth Apps is a 21-item self-report assessment of the acceptability (i.e., ease of use, interface and satisfaction, usefulness) of the mHealth application. Items are rated on a scale from 1 to 4 (possible range=21 to 84). Higher scores reflect greater acceptability of the mobile health app intervention.
Caregiver Qualitative Interview | 3 months post baseline
  These interviews will assess caregivers' perception of their relationship with their youth during their study involvement, as well as their feedback about whichever condition they were randomly assigned to, either the RAISE app or brochure.
Youth Qualitative Interview | After youth's release to the community within study period (estimated 2 years or less)
  Youth will be eligible to participate in a one-time qualitative interview if they have been released into the community while the study is being conducted. Youth interviews will assess their perceptions of support received from their caregiver, their caregiver's stress, and the role of their caregiver in facilitating connection to services.

CONTACTS AND LOCATIONS:
Overall Officials: Johanna B Folk, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Folk JB, McBride E, Nova S, Hurtado Y, Tolou-Shams M. Co-Design of the RAISE Mobile Health Intervention for and with Caregivers of Detained Youth. Res Child Adolesc Psychopathol. 2025 Dec;53(12):1813-1827. doi: 10.1007/s10802-025-01361-7. Epub 2025 Sep 22. PMID 40976844
- [Derived] Folk JB, Aguilera A, Chaplin TM, Tolou-Shams M. Stress Management Among Caregivers of Detained Youth: Protocol for Randomized Controlled Trial of the RAISE Web-Based mHealth App. JMIR Res Protoc. 2025 Jul 10;14:e67511. doi: 10.2196/67511. PMID 40638918